CLINICAL TRIAL: NCT03501290
Title: Compliance to Oral Nutritional Supplements (ONS) in Undernourished Frail Older Adults Living at Home.
Acronym: OFraDDom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Nutricia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/15/7814; 2015-A01870-49 (Other: ID-RCB)
Record Dates: First submitted 2017-11-13; First posted 2018-04-18 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Frail Elderly
Keywords: Frailty; Malnutrition; Older adults; Oral Nutritional Supplements; Compliance
MeSH Terms: conditions — Frailty; Malnutrition; Patient Compliance

STUDY DESIGN:
Intervention Model Description: All patients will be in one group, receiving the product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Nutritional Supplement Group (Other): All patients will be in one group, receiving the active product, Oral Nutritional Supplement with 'Fortimel® Protein supplementation'
  Interventions: Dietary Supplement: Fortimel® Protein supplementation

INTERVENTIONS:
Dietary Supplement: Fortimel® Protein supplementation — Patients are supposed to take Fortimel® Protein once daily during the study period. The prescription is one unit a day.
  First prescription of the study product will be done for one month. Prescription will be repeated for 2 additional months only after the patient's nutritional status and its global health status, as well as tolerability and compliance to the ONS, were re-assessed during the first follow-up visit at one month.

SUMMARY:
In this study, patients are supposed to take Fortimel® Protein, an Oral Nutritional Supplement (ONS) recommended in case of malnutrition once daily during the study period.

Three visits will be planned for each patient enrolled in the study (baseline visit, visits of follow-up at 4 weeks and 12 weeks). Phone calls will be regularly organized during one month or three months according to the duration of supplementation.

The primary purpose of the OFraDDom study is to assess the compliance with ONS (respect by the patient of the physician's prescription) at the end of the first month.

Data regarding the beneficial effects of ONS, or compliance with ONS in frail elderly population, are very limited. The study could complete knowledge about oral nutritional supplementation in the undernourished frail elderly people and help to demonstrate that oral nutritional supplements have benefits on nutritional status and physical performances in frail elderly people.

DETAILED DESCRIPTION:
For elderly with Protein Energy Malnutrition (PEM) or at nutritional risk, evidences support that Oral Nutritional Supplements (ONS) and dietary counselling can increase dietary intake and improve quality of life. However, data regarding the beneficial effects of ONS, or compliance with ONS in frail elderly population, are very limited. In their RCT, testing the effect of protein supplementation, Tieland and colleagues (7) showed an improvement of SPPB in frail older adults randomized to receive 15 g of supplemental protein daily for 24 weeks compared with the placebo group (p=0.02). Another recent RCT on the effect of a daily supplementation with protein and micronutrients for 12 weeks in 87 frail older adults (usual gait speed <0.6 m/s; MNA < 24) showed that Physical Functioning increased by 5.9% (1 point) in the intervention group, although no change was observed in the control group. SPPB remained stable in the intervention group, although it decreased by 12.5% (1 point) in controls (8).

In this study, patients are supposed to take Fortimel® Protein, an ONS recommended in case of malnutrition once daily during the study period.

Patients fulfilling eligibility criteria will be asked whether they are interested to participate in the study and receive Fortimel® protein. After informed consent, three visits will be planned for each patient enrolled in the study (baseline visit, visits of follow-up at 4 weeks and 12 weeks). Phone calls will be regularly organized during one month or three month according to the duration of supplementation to collect the compliance with ONS and coach patients.

First prescription of the study product will be done for one month. Prescription will be repeated for 2 additional months only after the patient's nutritional status and its global health status, as well as tolerability and compliance to the ONS, were re-assessed during the first follow-up visit at one month.

Data regarding the beneficial effects of ONS, or compliance with ONS in frail elderly population, are very limited. To complete knowledge about oral nutritional supplementation in the undernourished frail elderly people, study purpose is to assess Fortimel® Protein compliance to know if this supplementation is well accepted and what are factors which limit compliance. More, it could help to demonstrate that oral nutritional supplements have benefits on nutritional status and physical performances in frail elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* Pre-frail or frail as defined by Fried criteria: at least a low score on one of the following:

  * Weight loss
  * Exhaustion
  * Physical Activity
  * Walk time
  * Grip strength
* Undernutrition defined as at least one of the following criteria :

  * weight loss (≥ 5% in 1 month or ≥ 10% in 6 months),
  * BMI < 21 kg/m2
  * or global MNA <23.5
* Informed consent
* Willingness and ability to comply with the protocol, including:
* Participation in study visits
* Taking the study products every day
* Ability to perform test for physical functioning and frailty status
* Ability to understand and fill out questionnaires

Exclusion Criteria:

* Dependency or loss of autonomy: ADL<4
* Dementia
* MMSE ≤ <20 if study partner, MMSE<22 if loss of study partner
* Use of enteral nutrition
* Major depression: Geriatric Depression Scale >8
* Cancer with acute treatment (chemotherapy, radiotherapy)
* Allergy to cow milk proteins
* Galactosemia
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Fortimel® compliance | At the end of the first month : Day 30
  Fortimel® compliance as defined as the consumption of at least 75% of the prescribed volume of ONS.

SECONDARY OUTCOMES:
Fortimel® Compliance | Change at one and three months
  Fortimel® Compliance as defined as the consumption of at least 75% of the prescribed volume of ONS after 3 months supplementation,
Body weight evolution | Change at one and three months
  Body weight evolution measured during the follow up visits at one month and three months,
SPPB score | Change at one and three months
  Short Physical Performance Battery (SPPB) score (global score and each item)
MNA | Change at one and three months
  MNA scores evolution
ADL | Change at one and three months
  ADL scores evolution
Fragility : Fried criteria | Change at one and three months
  Fragility : Fried criteria evolution
EuroQoL | Change at one and three months
  EuroQoL scores evolution
Nutritional history intake | Change at one and three months
  Nutritional history intake evolution

CONTACTS AND LOCATIONS:
Overall Officials: Anne GHISOLFI, MD, Principal Investigator — Gérontopôle, CHU Toulouse
Locations (1):
- Toulouse University Hospital (CHU de Toulouse), Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided